CLINICAL TRIAL: NCT07183761
Title: A Randomized Controlled Trial Evaluating the Efficacy and Safety of Intramuscular Human Umbilical Cord Mesenchymal Stem Cell Therapy for Subjects With Moderate to Severe Diabetic Peripheral Neuropathy
Brief Title: A Randomized Controlled Trial on the Efficacy and Safety of Umbilical Cord Mesenchymal Stem Cell Therapy in Subjects With Moderate to Severe Diabetic Peripheral Neuropathy
Acronym: RELEASE-DPN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Min Long (Other)
Responsible Party: Sponsor-Investigator, Min Long, PhD, Associate Chief Physician, Associate Professor, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZD0509004-4.1
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Peripheral Neuropathy (DPN)
Keywords: Diabetic Peripheral Neuropathy; Mesenchymal Stem Cell Transplantation; Randomized Controlled Trial
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive three injections of hUC-MSCs (on Day 0, Day 7, and Day 28) while continuing conventional therapy.
  Interventions: Biological: Experimental Group; Drug: Conventional therapy group
- Control group (Active Comparator): The control group will receive conventional therapy only.
  Interventions: Drug: Conventional therapy group

INTERVENTIONS:
Biological: Experimental Group — On day 0, day 7, and day 28 after enrollment, the study subjects will receive intramuscular injections of hUC-MSCs suspension in normal saline into the medial and lateral muscle groups of both lower legs. Concurrently, all patients will continue to receive conventional therapy.
  Other Names: human umbilical cord mesenchymal stem cells (hUC-MSCs) injection
  Arms: Experimental group
Drug: Conventional therapy group — The conventional therapy include fundamental blood glucose management, basic treatment for diabetic neuropathy along with pain management therapy, as well as management of comorbidities and risk factors.
  Other Names: Conventional therapy

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of human umbilical cord mesenchymal stem cell (hUC-MSC) injection in the treatment of adults with moderate to severe diabetic peripheral neuropathy.

Researchers will compare hUC-MSCs injection combined with conventional therapy (experimental group) to conventional therapy alone (control group) to see if hUC-MSCs work to treat diabetic peripheral neuropathy.

The experimental group will receive three injections of hUC-MSCs (on Day 0, Day 7, and Day 28) while continuing conventional therapy, whereas the control group will receive conventional therapy only. Participants will undergo regular follow-ups for checkups and tests over a 24-week period. The primary endpoint of the study is the change in the Toronto Clinical Scoring System (TCSS) score at Week 24. Safety assessments will be conducted throughout the entire study period, with extended follow-up until Week 104 to evaluate long-term safety.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18-80 years;
2. Meeting the 2023 ADA diagnostic criteria for type 2 diabetes;
3. Presence of symptoms and signs of diabetic neuropathy in lower extremities:

   For symptomatic patients: At least one abnormal finding among ankle reflex, pinprick sensation, vibration sense, pressure perception, or temperature sensation, accompanied by clinical symptoms (e.g., symmetric lower limb numbness, pain, or tingling); For asymptomatic patients: At least two abnormal findings in the above five examinations;
4. Confirmed neurophysiological dysfunction:

   Reduced nerve conduction velocity (≥2 standard deviations) in at least one lower extremity nerve (common peroneal, posterior tibial, or deep peroneal nerve), with or without decreased amplitude;

   Moderate to severe neuropathy severity:
5. Toronto Clinical Scoring System (TCSS) score ≥9;
6. Inadequate response to conventional therapy: Persistent symptoms (reduction of TCSS score <2 points from baseline) despite ≥3 months of conventinal treatment;
7. Capacity to understand and voluntarily complete all study procedures and interventions, with signed informed consent.

Exclusion Criteria:

1. Non-diabetic neuropathy or pain conditions in lower limbs that may confound DPN assessment per investigator's judgment;
2. Poorly controlled diabetes (HbA1c >12%);
3. Severe hematological, hepatic, or renal dysfunction, meeting any of the following laboratory criteria:

   Hematology: Neutrophils <1.5×10⁹/L, platelets <90×10⁹/L, or hemoglobin <80 g/L; Liver function: ALT or AST >3× upper limit of normal (ULN), or total bilirubin >1.5× ULN; Renal function: eGFR <30 mL/min/1.73m² (calculated by MDRD formula) or requiring renal replacement therapy; Creatine kinase >2× ULN;
4. Known allergy to stem cells, stem cell-derived products, or components of stem cell preparations;
5. Current use of prohibited medications within 5 half-lives prior to enrollment (may be reconsidered after ≥5 half-lives washout);
6. Uncontrolled systemic diseases, including but not limited to: Severe uncontrolled systemic infections (bacterial, fungal, or viral); Severe autoimmune disorders; Hematological diseases; Heart failure (NYHA class ≥III);
7. Clinically significant arrhythmia on 12-lead ECG;
8. Conditions requiring amputation (e.g., severe diabetic foot or lower limb ulcers) that preclude local stem cell injection;
9. Other diseases unsuitable for trial participation (e.g., active malignancy, cognitive impairment, depression, or psychiatric disorders);
10. Participation in any interventional clinical trial within 3 months prior to screening;
11. Pregnancy, lactation, or planning pregnancy within 2 years;
12. Any other condition deemed by the investigator to compromise trial suitability.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Toronto Clinical Scoring System (TCSS) score | From enrollment to week 24 of the study period
  The TCSS is a method for assessing neurological function. It evaluates patients based on their symptoms, reflexes, and sensory test results to determine whether neurological impairment exists.
Incidence of stem cell-related adverse events | From enrollment to week 104 of the study period
  Safety endpoints
Incidence of stem cell-associated adverse reactions | From enrollment to week 104 of the study period
  Safety endpoints

SECONDARY OUTCOMES:
Nerve conduction velocity | From enrollment to week 24 of the study period
  Evaluated using electrophysiological studies to measure nerve conduction function
Quantitative Sensory Testing | From enrollment to week 24 of the study period
  Assess the participants' perception of temperature, vibration, and tactile sensations.
Pain Score | From enrollment to week 24 of the study period
  Assess the participants' pain score using visual analog scale (VAS).
Neuropathic pain | From enrollment to week 24 of the study period
  DN4 Neuropathic Pain Questionnaire
Health-related quality of life | From enrollment to week 24 of the study period
  EuroQol Five-Dimensional Five-Level Questionnaire (EQ-5D-5L)
Anxiety and Depression Scale | From enrollment to week 24 of the study period
  Hospital Anxiety and Depression Scale (HADS)

OTHER OUTCOMES:
Lower extremity blood flow velocity | From enrollment to week 24 of the study period
  Evaluated by lower limb vascular ultrasound
Microstructure of nerve fascicles | At enrollment and week 24 of the study period
  Evaluated by 7T MRI
Immune-inflammatory markers | At enrollment and week 24 of the study period
  Include erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), neutrophil-to-lymphocyte ratio (NLR), peripheral blood mononuclear cell subsets, and inflammation-related cytokines.
Status of lower extremity ulcers | At enrollment and week 104 of the study period
  The percentage of ulcer healing, along with the frequency and number of newly developed diabetic lower extremity ulcers

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided